CLINICAL TRIAL: NCT02761291
Title: Phase I Study of Cytolytic Viral Activation Therapy (CVAT) for Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Study of Cytolytic Viral Activation Therapy (CVAT) for Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-4750A
Record Dates: First submitted 2016-04-07; First posted 2016-05-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; EB virus; metastasis; recurrence; cytolytic viral activation therapy; gemcitabine; valproic acid; ganciclovir; valganciclovir
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections; Neoplasm Metastasis; Recurrence; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Gemcitabine; Valproic Acid; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine dose escalation (Experimental): In three combined drugs used in nasopharyngeal carcinoma, the valproic acid and valganciclovir administration will be followed by indication to find the maximum tolerance dose of gemcitabine.
  Interventions: Drug: Gemcitabine; Drug: Valproic acid; Drug: Valganciclovir

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administrated 600~1250 mg/m^2 intravenously according to the body surface area at day 1 and day 8 in a 28 day-treatment cycle. The treatment cycle of 28 days will be repeated maximum 6 times. The first dose level of gemcitabine will be started at 800 mg/m^2. If no subject suffered the dose limit toxicity, 1000 mg/m^2 and even 1250 mg/m^2 will be started by order. If subjects suffered the dose limit toxicity in 800 mg/m^2, the 600 mg/m^2 will be started.
  Other Names: Gemmis
Drug: Valproic acid — Valproic acid will be administrated orally by the fixed dose 12.5 mg/kg/day according to instructions from day 1 to day 14 in one treatment cycle. The treatment cycle of 28 days will be repeated maximum 6 times.
  Other Names: Depakine
Drug: Valganciclovir — Valganciclovir will be administrated orally by the fixed dose 1350 mg/day (creatinine clearance rate ≥ 60 mL/min) or 900 mg/day (creatinine clearance rate ≥ 40 mL/min and < 60 mL/min) from day 9 to day 15 in one treatment cycle. The treatment cycle of 28 days will be repeated maximum 6 times.
  Other Names: Valcyte

SUMMARY:
Nasopharyngeal carcinoma (NPC) is an Epstein-Barr virus(EBV) related malignancy and is an endemic disease in Southeast Asian countries. EBV had been identified as a therapeutic target in some EBV related cancer such as lymphoma and NPC. In cancer cell, EBV was in latent phase and expressed 8-11 genes for maintaining EBV proliferation. After switching to lytic phase, almost all the EBV encoding genes were expressed including thymidine kinase (TK) and some highly immunogenetic genes. These latent-lytic phase swifter included DNA methyltransferase inhibitors, various histone deacetylase (HDAC) inhibitors, radiotherapy and chemotherapy. Recently, combined chemotherapy and viral lytic therapy, cytolytic viral activation therapy (CVAT) had been shown some promising result in pilot study of NPC. In our patient derived xenograft (PDX) animal model drug sensitivity screening, gemcitabine (GEM) was shown to be the most effective drug. Furthermore, CVAT with GEM + Valproic acid (VPA) + ganciclovir (GCV) maintaining chemotherapy may benefit but reduce chemotherapy related side effect and prolonging treatment response duration. The following phase I clinical trial will be proposed to test the optimal combination of these drugs.

1. Number of patients: total 18 patients are needed
2. Inclusion criteria:(1) used as 2nd line regimen in recurrence/metastasis NPC patients with tissue proved of World Health Organization (WHO) type II or type III.(2) Performance status: eastern cooperative oncology group performance status (ECOG PS) ≤2.
3. Chemotherapy regimen: Gemcitabine (GEM, TTY) + Valproic acid (VPA, generic medicine) for viral activation + Valganciclovir (VGC, Roche) for antiviral medication
4. This treatment cycle of 28 days was repeated maximum 6 times. (Q4wks/cycle, max: 6 cycles)
5. Dosage:

(1) GEM: 600, 800, 1000, 1250 mg/m^2, D1 & D8, intravenously. (2) VPA 12.5 mg/kg/day D1~14, per os. (3) VGC (2-3) x 450 mg/day D9~15, per os. 6. Objectives:

1. primary: to find the best combination of these 3 drugs in recurrent/metastatic NPC patients.
2. second: to evaluate the response and disease control rate in this pilot study.

Key words: NPC, cytolytic viral activation therapy, gemcitabine, valproic acid, ganciclovir.

DETAILED DESCRIPTION:
1. Introduction to investigational treatment(s) and other study treatment(s)

   1.1 Overview of gemcitabine Gemcitabine (29,29-difluoro 29-deoxycytidine, dFdC) which developed from cytosine arabinoside (Ara-C) is an nucleoside analog used as chemotherapy. It was intended as an antiviral drug in initial, but preclinical testing showed that it killed leukemia cells and a spectrum of solid tumor in vitro. In cell, gemcitabine undergoes complex intracellular conversion to the active forms of nucleotides gemcitabine diphosphate (dFdCDP) and triphosphate (dFdCTP) that will influence DNA synthesis. dFdCTP competes with deoxycytidine triphosphate (dCTP) and dFdCDP is a potent inhibitor of ribonucleoside reductase (1). Gemcitabine is administered by the intravenous route with dose ranges from 0.6-1.2 g/m^2 of body surface area (2), and has been used in a broad spectrum cancer management including lung, breast, pancrease, and bladder (3).

   The toxic profile of gemcitabine was major in hematopoietic system especially neutropenia and thrombocytopenia (4). In NPC treatment, gemcitabine had been the focus of several reports, with interesting OR rates in the range of 23-48% and median progression-free survival (PFS) of between 3.6 and 5.1 months (5). In combination chemotherapy with cisplatin, the OR rate 42.7 to 73% had been reported and median PFS were 5.6 to 10.6 months (6). In combined with oxaliplatin, the OR rate was 56.1 % and median PFS was 9 months (6). In combined with vinorelbine, OR rate 36 to 37.7% had been reported and median PFS were 5.2 to 5.6 months. In multiple drugs combination with carboplatin, paclitaxel, 5-Fluoro-Uracil/LeucoVorin, high OR rate with 86% had been reported but with median PFS of 8 months (6). Still these trials were done in small series and lacking randomized large scale phase III trial.

   1.2 Valproic acid (VPA) Valproic acid (VPA), a branched short-chain fatty acid, is widely used in clinical as an antiepileptic drug and a mood stabilizer, primarily in the treatment of epilepsy, bipolar disorder, and prevention of migraine headaches (7). The antiepileptic properties of VPA have been attributed to inhibition of Gamma Amino Butyrate (GABA) trans aminobutyrate and of ion channels.

   VPA was recently classified among the Histone Deacetylase (HDAC) inhibitors, acting directly at the level of gene transcription by inhibiting histone deacetylation and making transcription sites more accessible. Chromatin is formed of DNA packaged in nucleosome structures. The condensed form of chromatin (heterochromatin) is inactive in terms of transcription whereas the decondensed form (euchromatin) corresponds to an active form. The histone acetylation leads to relaxation of the nucleosome structure, releasing the DNA and allowing transcription. Inhibition of histone deacetylases (HDACs) promotes decondensed chromatin formation, thereby promoting the expression of genes (7).

   Valproic acid (VPA), as a HDAC inhibitor, can specifically target at class I a, I b, and II a HDACs (8). VPA also down regulates expression of proteins essential for chromatin maintenance: Structural Maintenance of chromatin (SMC), DNA methyl transferase-1 (DNMT1), and heterochromatin protein-1 (HP1) (9). VPA had been shown to induce histone 3 methylation which would increase transcriptional activity (8). VPA had been shown some anticancer effect, major through its HDAC inhibitor, in single agent or combined with other anticancer medication including myeloid and lymphoid malignancies, breast cancer, prostate cancer, and NPC (10-13) Long-term VPA treatment may cause central nervous system (CNS) dysfunction, liver toxicity, and coagulopathy including thrombocytopenia and platelet dysfunction (7).

   1.3 Ganciclovir (GCV) and Valganciclovir (VGC) GCV was an antiviral agent had been used in treatment or prophylaxis of cytomegalovirus infection in solid organ transplantation recipients or bone marrow transplantation (14). GCV is a synthetic analogue of 2'-deoxy-guanosine and can be phosphorylated to ganciclovir triphosphate, a competitive inhibitor of deoxyguanosine triphosphate (dGTP) incorporation into DNA and preferentially inhibits viral DNA polymerases more than cellular DNA polymerases, by viral and cell kinase. In addition, ganciclovir triphosphate serves as a poor substrate for chain elongation, thereby disrupting viral DNA synthesis by a second route (15).

   VGC, a valyl ester prodrug of GCV, had a high oral bioavailability of about 60% with similar efficacy of GCV in management of cytomegalovirus infection (16). The most common side effect of IV GCV is fever and leukopenia (16).

   1.4 Combination of GEM, VPA and GCV in NPC treatment In EBV-related malignancy, antiviral drugs exhibit no direct effect on cancer cell except when used combined with epigenetically active agents (17, 18). Recently, Wildeman et al, had shown some efficacy by combining chemotherapy of GEM with VPA and GCV in control of locally advanced/metastatic NPC patients (13). In this article, both GEM and VPA could shift EBV from latent phase into lytic phase and had synergetic effect when combined used. Further adding GCV in this regimen could suppress virion formation. The combination therapy had been tested in three locally advanced/metastatic NPC patients showing promising results with tumor regressing/stable in image and plasma EBV DNA load monitoring with few side effects Similar manageable side effects of these three drugs combined treatment were also proved by Stoker et al (19). These results encouraged us to develop a more practical regimen in this trial.
2. Test products, dosage, and mode of administration:

2.1. Chemotherapy regimen: Gemcitabine (Gemmis injection，200 mg) (GEM, TTY) + Valproic acid (Depakine gastro-resistant tablet，200 mg) (VPA, Sanofi) for viral activation + Valganciclovir (Valcyte film-coated tablets，450 mg) (VGC, Roche) for antiviral medication

2.2. Dosage GEM: 600~1250 mg/m^2, D1 & D8, intravenously. VPA: 12.5 mg/kg/day D1~14, per os. VGC: (2~3) x 450mg/day D9~15, per os.

1. This treatment cycle of 28 days will be repeated maximum 6 times. (Q4wks/cycle, max: 6 cycles)
2. Four dosage of GEM combined with fixed dosage of VPA and VGC will be tested
3. The rationale of seven days treatment duration of VGC come from (A) 7 days treatment duration of valacyclovir in herpes zoster in immunocompetent patients (20) (B) overlap side effect of myelosuppression between GEM and VGC(13).
4. Efficient dose intensity chemotherapy (gemcitabine) is essential in this three combined drugs regimen (21) and this trial will be started with dose level 0 (Gemcitabine 800 mg/m^2)

2.3. Concomitant treatment

2.3.1 Permitted: The related treatment for relieve symptoms caused from tumor.

2.3.2 Prohibited:

1. Radiation therapy, operation, and other chemotherapy for eradicating tumor
2. Valganciclovir concomitant with Imipenem-cilastatin could result in convulsion; with zidovudine could result in neutropenia; with Probenecid would increase toxicity of ganciclovir
3. Co-administration of valproate with amitryptyline/nortryptyline, and warfarin need to be adjusted if necessary
4. Co-administration of valganciclovir with didanosine, Mycophenolate mofetil, and bone marrow suppression drugs (e.g., dapsone, pentamidine, flucytosine, vincristine, vinblastine, adriamycin, amphotericin B, nucleoside analogues, hydroxyurea) would need to be monitored more seriously because of their toxicity might increase
5. All other drugs prohibited co-administration with valproic acid absolutely

3. Duration of treatment: This treatment cycle of 28 days will be repeated maximum 6 times. (Q4wks/cycle, max: 6 cycles) A standard 3 + 3 phase I dose escalation study design was used (22). A minimum of three evaluable patients were to be treated at each dose level. According to Worst Toxicity CTCAE v4.03 Grade and FDA indication of gemcitabine, the dose limiting toxicity (DLT) of this trial was determined in the first treatment cycle.

In the absence of DLT, patients were enrolled in the next dose level. If 1 of three patients had a DLT, the cohort was expanded to include six patients. If ≥2 patients experienced DLT, maximum tolerated dose (MTD) was exceeded and further enrollment at that dose level was stopped. MTD was defined as the highest dose level at which ≤1 of 6 patients experienced a DLT. Only DLT that occurred during the first treatment cycle were used to determine the MTD.

4. Patient examination and re-evaluation: Laboratory data of complete blood count (CBC)/differential count (DC), creatinine, alanine aminotransferase (ALT) will be routine checked every weeks during the first 3 treatment cycles. During all treatment courses, if grade 4 neutropenia or grade 4 thrombocytopenia attacked, the laboratory will be checked every 3 days until recovered to pre-treatment baseline. Around 70% responsive and stable cases could be enrolled in the 4th treatment cycle will be routine checked the laboratory data before gemcitabine administration. Plasma EBV DNA copies number will be monitored before each cycle treatment. Systemic re-evaluation will be performed after every three cycles treatment. Re-evaluation including physical examination, image studies including CT/MRI for head and neck area, chest x-ray, abdominal echo, and Gallium whole body tumor scan, and blood exam including complete CBC count, biochemical profile, and plasma EBV DNA copies number.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand and willingness to sign a written informed consent document
2. Identified as recurrent nasopharyngeal carcinoma or distant metastases of male or female subjects who had failed in 1st line therapy including radiotherapy, not suitable for radiotherapy or unwilling to receive radiotherapy, 1st line chemotherapy excluding gemcitabine, and no curative treatment options
3. Biopsy confirmed belong to World Health Organization classification of nasopharyngeal carcinoma type II or type III
4. Men and women between aged 20 to 80 years of age; female patients with childbearing potential will routinely consult obstetric doctor for contraception and need to have contraception at least 6 months after finished this trial
5. Adequate internal organs including liver, kidney and bone marrow function

   * white blood cell count of >3,000/µL; platelet count of ≥100,000/µL; absolute neutrophil count >1,500/µL
   * total bilirubin <2.0 mg/dL, aspartate aminotransferase (AST), alanine transaminase(ALT) <2.5x upper limit of normal range (ULN)
   * serum creatinine <2.0 mg/dL
6. The daily performance status ECOG ≤ 2 points

Exclusion Criteria:

1. Pregnancy or breast-feeding women, and plans within six months of pregnancy
2. Contraindication to Gemmis injection, Depakine gastro-resistant tablet, and Valcyte film-coated tablets, including:

   * Allergy to Gemmis injection, Depakine gastro-resistant tablet, Valcyte film-coated tablets, and other similar drugs
   * Patients with hepatic B or C, patients with human immunodeficiency virus, or viral related disease receiving anti-viral treatment
   * Acute or chronic hepatitis not related to NPC with liver metastasis
   * Using drugs which ineligible combination with valproic acid, including mefloquine, St.-John's-Wort, lamotrigine, Topiramate, quetiapine, cyclosporin, hepatic enzyme-inducing drugs (e.g., phenytoin, carbamazepine phenobarbital, primidone, rifampin), enzyme inhibitors (e.g., felbamate), aspirin, cimetidine, erythromycin, carbapenem (e.g., Panipenem, Aztreonam, Imipenem, Meropenem), diazepam, ethosuximide, lamotrigine, phenytoin, nimodipine
3. With insomnia, anxiety or spiritual concerns, or are receiving mental illness treatment
4. Has been diagnosed with a second cancer, except to basal cell carcinoma
5. Patients unsuitable to this trial, including:

   * Patients with significant disease
   * PI evaluated with high risk group patients
   * Patients not recovered from previous anti-cancer treatment
   * Recent major surgery
6. Patients with creatinine clearance rate <40 ml/min

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants suffered dose limiting toxicity (DLT) that are related to this treatment | The first treatment cycle (1~28 days approximately)
  According to Worst Toxicity CTCAE v4.03 Grade and FDA indication of gemcitabine, the dose limiting toxicity (DLT) of this trial was determined in the first treatment cycle and DLTs were defined as ≥1 of the following effects attributable to the study drug and requiring discontinuation or a significant dose reduction in the study drug(s):
  1. ≥Grade 4 neutropenia >5 days;
  2. ≥Grade 4 thrombopenia lasting ≥7 days;
  3. ≥Grade 3 anemia;
  4. ≥Grade 3 neutropenic fever with a single temperature of >38.3 degree C or a sustained temperature of ≥ 38 degree C for more than one hour;
  5. any ≥Grade 3 non-hematologic toxicity with exception of nausea and vomiting, alopecia, drug-related fever;
  6. ≥Grade 3 serum creatinine;
  7. bone marrow and renal function didn't recover to CTCAE Grade ≤ 1 of baseline at the Day 1 of the 2nd treatment course, the treatment can be postponed less than 2 weeks. DLT was recognized when the delayed duration was more than 2 weeks.

SECONDARY OUTCOMES:
Safety and tolerability assessed by adverse events, serious adverse events | 3~6 months
Overall Response Rate (ORR), according to RECIST criteria, assessed by CT/MRI for head and neck area/chest x-ray/abdominal echo/Gallium whole body tumor scan | 3~6 months in treatment, and 3~6 months in followed-up
EB virus DNA load in plasma | 3~6 months in treatment, and 3~6 months in followed-up
  The plasma EB virus DNA load will be check by real-time quantitative polymerase chain reaction (PCR). These data will be collected every months when subjects enter this trial and finish their final treatment cycle one weeks, 3 months, and/or 6 months later. These data will be used to supplementary data for tumor status assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Lung Hsu, Physican, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang-Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mini E, Nobili S, Caciagli B, Landini I, Mazzei T. Cellular pharmacology of gemcitabine. Ann Oncol. 2006 May;17 Suppl 5:v7-12. doi: 10.1093/annonc/mdj941. PMID 16807468
- [Background] Wang LR, Liu J, Huang MZ, Xu N. Comparison of pharmacokinetics, efficacy and toxicity profile of gemcitabine using two different administration regimens in Chinese patients with non-small-cell lung cancer. J Zhejiang Univ Sci B. 2007 May;8(5):307-13. doi: 10.1631/jzus.2007.B0307. PMID 17542057
- [Background] Noble S, Goa KL. Gemcitabine. A review of its pharmacology and clinical potential in non-small cell lung cancer and pancreatic cancer. Drugs. 1997 Sep;54(3):447-72. doi: 10.2165/00003495-199754030-00009. PMID 9279506
- [Background] Natale R. A ten-year review of progress in the treatment of non-small-cell lung cancer with gemcitabine. Lung Cancer. 2005 Oct;50 Suppl 1:S2-4. doi: 10.1016/s0169-5002(05)81549-1. PMID 16291427
- [Background] Bensouda Y, Kaikani W, Ahbeddou N, Rahhali R, Jabri M, Mrabti H, Boussen H, Errihani H. Treatment for metastatic nasopharyngeal carcinoma. Eur Ann Otorhinolaryngol Head Neck Dis. 2011 Apr;128(2):79-85. doi: 10.1016/j.anorl.2010.10.003. Epub 2010 Dec 21. PMID 21177151
- [Background] Xu T, Tang J, Gu M, Liu L, Wei W, Yang H. Recurrent nasopharyngeal carcinoma: a clinical dilemma and challenge. Curr Oncol. 2013 Oct;20(5):e406-19. doi: 10.3747/co.20.1456. PMID 24155638
- [Background] Chateauvieux S, Morceau F, Dicato M, Diederich M. Molecular and therapeutic potential and toxicity of valproic acid. J Biomed Biotechnol. 2010;2010:479364. doi: 10.1155/2010/479364. Epub 2010 Jul 29. PMID 20798865
- [Background] Bradbury CA, Khanim FL, Hayden R, Bunce CM, White DA, Drayson MT, Craddock C, Turner BM. Histone deacetylases in acute myeloid leukaemia show a distinctive pattern of expression that changes selectively in response to deacetylase inhibitors. Leukemia. 2005 Oct;19(10):1751-9. doi: 10.1038/sj.leu.2403910. PMID 16121216
- [Background] Marchion DC, Bicaku E, Daud AI, Sullivan DM, Munster PN. Valproic acid alters chromatin structure by regulation of chromatin modulation proteins. Cancer Res. 2005 May 1;65(9):3815-22. doi: 10.1158/0008-5472.CAN-04-2478. PMID 15867379
- [Background] Kuendgen A, Strupp C, Aivado M, Bernhardt A, Hildebrandt B, Haas R, Germing U, Gattermann N. Treatment of myelodysplastic syndromes with valproic acid alone or in combination with all-trans retinoic acid. Blood. 2004 Sep 1;104(5):1266-9. doi: 10.1182/blood-2003-12-4333. Epub 2004 May 20. PMID 15155466
- [Background] Ma BB, Chan AT. Recent perspectives in the role of chemotherapy in the management of advanced nasopharyngeal carcinoma. Cancer. 2005 Jan 1;103(1):22-31. doi: 10.1002/cncr.20768. PMID 15565580
- [Background] Duenas-Gonzalez A, Candelaria M, Perez-Plascencia C, Perez-Cardenas E, de la Cruz-Hernandez E, Herrera LA. Valproic acid as epigenetic cancer drug: preclinical, clinical and transcriptional effects on solid tumors. Cancer Treat Rev. 2008 May;34(3):206-22. doi: 10.1016/j.ctrv.2007.11.003. Epub 2008 Jan 15. PMID 18226465
- [Background] Wildeman MA, Novalic Z, Verkuijlen SA, Juwana H, Huitema AD, Tan IB, Middeldorp JM, de Boer JP, Greijer AE. Cytolytic virus activation therapy for Epstein-Barr virus-driven tumors. Clin Cancer Res. 2012 Sep 15;18(18):5061-70. doi: 10.1158/1078-0432.CCR-12-0574. Epub 2012 Jul 3. PMID 22761471
- [Background] Vaziri S, Pezhman Z, Sayyad B, Mansouri F, Janbakhsh A, Afsharian M, Najafi F. Efficacy of valganciclovir and ganciclovir for cytomegalovirus disease in solid organ transplants: A meta-analysis. J Res Med Sci. 2014 Dec;19(12):1185-92. PMID 25709661
- [Background] Noble S, Faulds D. Ganciclovir. An update of its use in the prevention of cytomegalovirus infection and disease in transplant recipients. Drugs. 1998 Jul;56(1):115-46. doi: 10.2165/00003495-199856010-00012. PMID 9664203
- [Background] Len O, Gavalda J, Aguado JM, Borrell N, Cervera C, Cisneros JM, Cuervas-Mons V, Gurgui M, Martin-Davila P, Montejo M, Munoz P, Bou G, Carratala J, Torre-Cisneros J, Pahissa A; RESITRA. Valganciclovir as treatment for cytomegalovirus disease in solid organ transplant recipients. Clin Infect Dis. 2008 Jan 1;46(1):20-7. doi: 10.1086/523590. PMID 18171208
- [Background] Ghosh SK, Perrine SP, Williams RM, Faller DV. Histone deacetylase inhibitors are potent inducers of gene expression in latent EBV and sensitize lymphoma cells to nucleoside antiviral agents. Blood. 2012 Jan 26;119(4):1008-17. doi: 10.1182/blood-2011-06-362434. Epub 2011 Dec 7. PMID 22160379
- [Background] Olson D, Gulley ML, Tang W, Wokocha C, Mechanic O, Hosseinipour M, Gold SH, Nguluwe N, Mwansambo C, Shores C. Phase I clinical trial of valacyclovir and standard of care cyclophosphamide in children with endemic Burkitt lymphoma in Malawi. Clin Lymphoma Myeloma Leuk. 2013 Apr;13(2):112-8. doi: 10.1016/j.clml.2012.11.003. Epub 2012 Dec 20. PMID 23260601
- [Background] Stoker SD, Novalic Z, Wildeman MA, Huitema AD, Verkuijlen SA, Juwana H, Greijer AE, Tan IB, Middeldorp JM, de Boer JP. Epstein-Barr virus-targeted therapy in nasopharyngeal carcinoma. J Cancer Res Clin Oncol. 2015 Oct;141(10):1845-57. doi: 10.1007/s00432-015-1969-3. Epub 2015 Apr 29. PMID 25920375
- [Background] Gnann Jr. JW. Antiviral therapy of varicella-zoster virus infections. In: Arvin A, Campadelli-Fiume G, Mocarski E, Moore PS, Roizman B, Whitley R, Yamanishi K, editors. Human Herpesviruses: Biology, Therapy, and Immunoprophylaxis. Cambridge: Cambridge University Press; 2007. Chapter 65. Available from http://www.ncbi.nlm.nih.gov/books/NBK47401/ PMID 21348091
- [Background] Mascarenhas L, Malogolowkin M, Armenian SH, Sposto R, Venkatramani R. A phase I study of oxaliplatin and doxorubicin in pediatric patients with relapsed or refractory extracranial non-hematopoietic solid tumors. Pediatr Blood Cancer. 2013 Jul;60(7):1103-7. doi: 10.1002/pbc.24471. Epub 2013 Jan 17. PMID 23335436
- [Result] Hsu CL, Kuo YC, Huang Y, Huang YC, Lui KW, Chang KP, Lin TL, Fan HC, Lin AC, Hsieh CH, Lee LY, Wang HM, Li HP, Chang YS. Application of a patient-derived xenograft model in cytolytic viral activation therapy for nasopharyngeal carcinoma. Oncotarget. 2015 Oct 13;6(31):31323-34. doi: 10.18632/oncotarget.5544. PMID 26416517